CLINICAL TRIAL: NCT00056277
Title: Double Blind Placebo Controlled Study of Lamictal in Acute Bipolar Depression
Brief Title: Bipolar Disorder Study for Men and Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCA30924
Record Dates: First submitted 2003-03-10; First posted 2003-03-11 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Drug: lamotrigine

INTERVENTIONS:
Drug: lamotrigine

SUMMARY:
A Placebo Controlled Study Evaluating Efficacy and Safety of Medication in Patients with Bipolar Disorder

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide written and informed consent
* Diagnosis of Bipolar I Disorder and currently depressed for minimum of the previous 8 weeks
* Patients must have been hospitalized for mood disorder or incarceration with or without formal charges as the result of mania related behavior

Exclusion Criteria:

* Patients must not be suicidal
* Patients must not have a history or non-response to antidepressant treatment
* Patients must not have a clinical history of substance dependence in the past year or abuse within the 4 weeks prior to study entry
* Patients must not have had epilepsy or hypothyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2003-02-27; Primary Completion 2005-08-01 (Actual); Study Completion 2005-12-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline scores at Week 8 for the Montgomery-Asberg Depression Rating Scale (MADRS) | 8 Weeks

SECONDARY OUTCOMES:
Change from baseline scores at Week 8 for the Hamilton Depression Rating Scale (HAMD-17, HAMD-31, Bech Melancholia Scale (BMS), and HAMD - Item 1), Clinical Global Impressions of Severity (CGI-S) and Improvement (CGI-I). | 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (20):
- United States (20):
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Terre Haute, Indiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Princeton, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Pleasantville, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Brecksville, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Brown Deer, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Hashimoto Y, Kotake K, Watanabe N, Fujiwara T, Sakamoto S. Lamotrigine in the maintenance treatment of bipolar disorder. Cochrane Database Syst Rev. 2021 Sep 15;9(9):CD013575. doi: 10.1002/14651858.CD013575.pub2. PMID 34523118
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: SCA30924 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SCA30924 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SCA30924 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SCA30924 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SCA30924 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SCA30924 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SCA30924 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register